CLINICAL TRIAL: NCT01074983
Title: Prevalence of Pre-hospital Hypoxemia in Trauma Patients: Do Trauma Patients Need Oxygen?
Brief Title: Pre-hospital Hypoxemia in Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Jason McMullan, Associate Clinical Professor, University of Cincinnati
Other Study IDs: FA8650-05-2-6518-661150
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Trauma
Keywords: Prehospital, Oxygen, Trauma, Hypoxemia
MeSH Terms: conditions — Wounds and Injuries; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Written standard of care
- Usual practice pattern

SUMMARY:
The intent of this study is to describe the proportion of trauma patients requiring oxygen before hospital arrival, the amount of oxygen they require, and whether or not the oxygen is beneficial to outcomes.

DETAILED DESCRIPTION:
Trauma patients in the United States frequently receive high-flow high-concentration supplemental oxygen in the pre-hospital setting, yet their physiologic need is rarely known. Providing oxygen to everyone regardless of need may seem straightforward, but the practice has extensive implications in logistically challenging areas such as a combat arena or mass casualty event, and is not supported by care guidelines. Indeed, too much oxygen can be harmful for some patients.1, 2 If it is the case, that not all trauma patients require oxygen, this would decrease the logistical burden of providing oxygen in the pre-hospital environment. No study has yet been performed that describes the proportion of patients requiring oxygen, the amount of oxygen they require, and whether or not oxygen is beneficial to outcomes. This prospective observational cohort investigation aims to bridge the knowledge gap surrounding the need and possible benefits or harms arising from oxygen therapy. In our Emergency Medical Services (EMS) systems, the written standard of care is to provide oxygen only to maintain oxygen saturation at 95% or when hemorrhagic shock or traumatic brain injury are suspected.3 We will observe patterns of oxygen treatment and outcome for patients treated according to this written standard of care, and compare this to the treatment and outcomes for patients transported by EMS units who continue their usual practice pattern.

Specifically, we aim to:

1. Identify the proportion of trauma patients who are hypoxemic or who have traumatic brain injury or hemorrhagic shock at the time of initial EMS contact
2. Identify the proportion of trauma patients who develop hypoxemia or hemorrhagic shock while in the pre-hospital setting
3. Identify differences in clinically important outcomes associated with treatments driven by written standard of care compared with the usual practice pattern of EMS units. These outcomes include requirement for advanced airway management, hospital and intensive care unit lengths of stay, and disposition (including in-hospital and 30-day mortality)
4. Determine the amount of oxygen (Liters per minute) required to reverse hypoxemia

ELIGIBILITY:
Inclusion Criteria:

* acute traumatic injury
* transported directly to study hospital
* meets at least one trauma consult/trauma stat criteria

Exclusion Criteria:

* lack of continuous peripheral pulse oximetry data
* age <18 years
* on prescribed home oxygen therapy prior to trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients arriving at a Level 1 Trauma Center by designated EMS units
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of trauma patients who are hypoxemic or who have traumatic brain injury or hemorrhagic shock at the time of initial emergency medical services (EMS) contact | At enrollment

SECONDARY OUTCOMES:
Proportion of trauma patients who develop hypoxemia or hemorrhagic shock while in the pre-hospital setting | at enrollment
Amount of oxygen required to correct hypoxemia | at enrollment
Clinically important outcomes associated with treatments driven by written standard of care compared with the usual practice pattern of EMS units | at study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jason T McMullan, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States